CLINICAL TRIAL: NCT00771160
Title: MK0476 Phase III Long-term Study -Perennial Allergic Rhinitis-
Brief Title: MK0476 Study in Adult Patients With Perennial Allergic Rhinitis (0476-397)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0476-397; 2008_553
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic | interventions — montelukast

ARMS (2):
- 1 (Experimental): MK0476 5mg
  Interventions: Drug: montelukast sodium
- 2 (Experimental): MK0476 10mg
  Interventions: Drug: montelukast sodium

INTERVENTIONS:
Drug: montelukast sodium — Arm 1: montelukast tablet 5 mg, QD. Treatment period is 12-weeks. Arm 2: montelukast tablet 10 mg, QD. Treatment period is 12-weeks.
  Other Names: Singulair

SUMMARY:
A clinical study evaluates the efficacy and safety of MK0476 in adult patients with Perennial Allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients With Perennial Allergic Rhinitis

Exclusion Criteria:

* Patients Who Have Nasal Diseases (E.G., Nasal Polyp, Septonasal Arcuation, Hypertrophic Rhinitis), Upper Respiratory Infection, Sinusitis, Infectious Rhinitis And Those Disease Severe Enough To Interfere With Assessment Of Effectiveness
* Patients Who Have Rhinitis Medicamentosa, Or Nonallergic Rhinitis (E.G., Vasomotor Rhinitis, Eosinophilia Rhinitis)
* Patient Has A Disease Of The Cardiovascular, Hepatic, Renal, Hematologic Systems, Or Other Severe Disease

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-09; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Any clinical or laboratory adverse experience | 12 weeks

SECONDARY OUTCOMES:
The daily mean of the composite nasal symptoms score at each of biweekly visits during the treatment period (average over the previous 2 weeks) or at time of termination | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC